CLINICAL TRIAL: NCT00110019
Title: A Double-Blind, Randomized, Placebo-Controlled Phase III Trial of Carboplatin, Paclitaxel and Sorafenib Versus Carboplatin, Paclitaxel and Placebo in Patients With Unresectable Locally Advanced or Stage IV Melanoma
Brief Title: Carboplatin and Paclitaxel With or Without Sorafenib Tosylate in Treating Patients With Stage III or Stage IV Melanoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02978; NCI-2012-02978 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E2603 (Other: ECOG-ACRIN Cancer Research Group); E2603 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-07

CONDITIONS: Mucosal Melanoma; Recurrent Melanoma; Stage IIIA Skin Melanoma; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — Carboplatin; Paclitaxel; Taxes; Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (paclitaxel, carboplatin, sorafenib tosylate) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Patients also receive sorafenib tosylate PO BID (approximately every 12 hours) on days 2-19.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study; Drug: Sorafenib Tosylate
- Arm II (carboplatin, paclitaxel, placebo) (Active Comparator): Patients receive paclitaxel and carboplatin as in Arm I. Patients also receive placebo PO BID (approximately every 12 hours) on days 2-19.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study; Other: Placebo

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (carboplatin, paclitaxel, placebo)
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
  Arms: Arm I (paclitaxel, carboplatin, sorafenib tosylate)

SUMMARY:
This randomized phase III trial studies carboplatin, paclitaxel, and sorafenib tosylate to see how well they work compared to carboplatin and paclitaxel in treating patients with stage III or stage IV melanoma that cannot be removed by surgery. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether giving carboplatin and paclitaxel together with sorafenib tosylate is more effective than carboplatin and paclitaxel in treating melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the overall survival of patients with unresectable stage III or stage IV melanoma treated with carboplatin, paclitaxel and placebo versus carboplatin, paclitaxel and sorafenib (sorafenib tosylate).

II. To compare progression-free survival, response rate, and safety of patients with unresectable stage III or stage IV melanoma treated with carboplatin, paclitaxel and placebo versus carboplatin, paclitaxel and sorafenib.

III. To analyze the pharmacokinetic and pharmacogenetic properties of sorafenib including angiogenesis, monooxygenases polymorphisms and multidrug resistance (MDR).

IV. To assess the association of expression markers in the patient tumor with clinical outcome.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes on day 1. Patients also receive sorafenib tosylate orally (PO) twice daily (BID) (approximately every 12 hours) on days 2-19.

Arm II: Patients receive paclitaxel and carboplatin as in Arm I. Patients also receive placebo PO BID (approximately every 12 hours) on days 2-19.

In both arms, treatment repeats every 21 days for 10 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease or who achieve a partial response or complete response may continue to receive sorafenib tosylate or placebo alone BID (approximately every 12 hours) on days 1-21. Courses with sorafenib tosylate or placebo repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed melanoma that is metastatic or unresectable; patients must have a history of cutaneous, mucosal or unknown primary site
* Patients who have received prior systemic cytotoxic chemotherapy for treatment of melanoma are ineligible; the following groups are eligible with regard to prior systemic therapy either in the adjuvant or metastatic disease setting:

  * No prior therapy
  * Immunotherapy consisting of interferon, interleukin-2, granulocyte macrophage colony-stimulating factor (GM-CSF) or vaccine
  * One prior investigational therapy (cannot be chemotherapy or an inhibitor of rat sarcoma [Ras], serine/threonine kinase [Raf], or mitogen-activated protein kinase kinase [MEK])

    * NOTE: Chemotherapy given via isolated limb perfusion is allowed
* Prior radiation therapy is allowed; however, if radiation has been administered to a lesion, there must be radiographic evidence of progression of that lesion in order for that lesion to constitute measurable disease or to be included in the measured target lesions
* All sites of disease must be evaluated within 4 weeks of registration; patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* White blood count >= 3,000/mm^3
* Absolute granulocyte count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Serum creatinine =< 2.0 x upper limit of normal (ULN) or serum creatinine clearance (CrCl) >= 40 ml/min (neither drug is cleared by the kidney)
* Total bilirubin =< 1.5 x ULN (< 3.0 x ULN in the presence of Gilbert's disease)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN (=< 5.0 ULN in the presence of liver metastases)
* International normalized ratio (INR) =< 1.5 and a partial thromboplastin time (PTT) within normal limits (patients who are on therapeutic anticoagulation with warfarin should have documentation of a normal prothrombin time [PT]/PTT prior to initiating that therapy)
* Patients must not have ocular melanoma
* Patients must have discontinued immunotherapy or radiation therapy at least 4 weeks prior to initiation of treatment and recovered from adverse events due to those agents
* Patients must not receive any other investigational agents during the period on study or the four weeks prior to initiation of treatment
* Patients must not have a history or clinical evidence of brain metastasis; patients must be evaluated with a head magnetic resonance imaging (MRI) within 4 weeks prior to enrollment
* Patients must not have other current malignancies, other than basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast; patients with other malignancies are eligible if they have been continuously disease-free for >= 5 years prior to the time of randomization
* Patients must not have any evidence of bleeding diathesis
* Patients must not have a serious intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics, clinically significant cardiovascular disease (e.g. uncontrolled hypertension, myocardial infarction, unstable angina), New York Heart Association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or grade II or greater peripheral vascular disease within 1 year prior to study entry, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not be taking cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or phenobarbital), rifampin or St. John's Wort
* Women must not be pregnant or breast-feeding
* All females of childbearing potential must have a blood test or urine study within 4 weeks prior to registration to rule out pregnancy
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant while participating in this study, she should inform her treating physician immediately; if a man impregnates a woman while participating in this study, he should inform his treating physician immediately as well
* Human immunodeficiency virus (HIV)-positive patients are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2005-06; Primary Completion 2011-01 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Flaherty, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (219):
- United States (218):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Marin Cancer Care Inc, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Bay Area Tumor Institute, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Veterans Administration-San Diego Medical Center, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Santa Rosa Memorial Hospital, Sana Rosa, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Southwest Florida Regional Medical Center, Fort Meyers, Florida
  - University of Florida, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - IU Health Bloomington, Bloomington, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Central Maine Medical Center, Lewiston, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Commonwealth Hematology Oncology PC-Worcester, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Unity Hospital, Fridley, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hackensack University Medical CCOP, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Laura and Issac Perlmutter Cancer Center at NYU Langone, New York, New York
  - MidHudson Regional Hospital of Westchester Medical Center, Poughkeepsie, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Wooster Specialty Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Western Oncology Research Consortium, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, DuBois, Pennsylvania
  - PinnacleHealth Cancer Center-Community Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Kent County Hospital, Warwick, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - East Tennessee Baptist Hospital-Mercy Health Partners, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Vermont College of Medicine, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes, Elkhorn, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Sydney West Area Health Service-Westmead Hospital, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] Flaherty KT, Lee SJ, Zhao F, Schuchter LM, Flaherty L, Kefford R, Atkins MB, Leming P, Kirkwood JM. Phase III trial of carboplatin and paclitaxel with or without sorafenib in metastatic melanoma. J Clin Oncol. 2013 Jan 20;31(3):373-9. doi: 10.1200/JCO.2012.42.1529. Epub 2012 Dec 17. PMID 23248256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on June 23, 2005, and terminated on April 22, 2008 with the final accrual of 823 patients. Most of patients were accrued through Eastern Cooperative Oncology Group (ECOG), Cancer and Leukemia Group B (CALGB), and Southwest Oncology Group (SWOG). Other Clinical Trials Cooperative Groups also participated.
Groups:
- Arm I (Carboplatin+Paclitaxel+Sorafenib): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Patients also receive oral sorafenib twice daily on days 2-19.
- Arm II (Carboplatin+Paclitaxel): Patients receive paclitaxel and carboplatin as in arm I. Patients also receive oral placebo twice daily on days 2-19.
Period: Overall Study
Arm/Group | Arm I (Carboplatin+Paclitaxel+Sorafenib) | Arm II (Carboplatin+Paclitaxel)
Started | 410 | 413
Eligible | 395 | 398
Treated | 393 | 397
Completed | 4 | 0
Not Completed | 406 | 413
Not completed — Lack of Efficacy | 253 | 285
Not completed — Adverse Event | 61 | 40
Not completed — Death | 13 | 15
Not completed — Withdrawal by Subject | 21 | 9
Not completed — alternative therapy | 5 | 1
Not completed — complicating disease | 1 | 1
Not completed — symptom deterioration | 13 | 16
Not completed — Not start protocol therapy | 17 | 16
Not completed — other reasons | 22 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Carboplatin+Paclitaxel+Sorafenib) | Arm II (Carboplatin+Paclitaxel) | Total
Number analyzed (Participants) | 410 | 413 | 823
Age, Continuous [Median (Full Range); unit: years] | 60 [19 to 86] | 58 [18 to 84] | 59 [18 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 162 | 302
  Male | 270 | 251 | 521

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as time from study entry to death from any cause. The comparison of overall survival was conducted in intention-to-treat population.
Time Frame: Survival was assessed every 3 months if patient is < 2 years from study entry. Every 6 months is patient is 2-5 years from study entry.
Population: Intention-to-treat population, n=823
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm I (Carboplatin + Paclitaxel + Sorafenib): Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes on day 1. Patients also receive oral sorafenib twice daily on days 2-19.
- Arm II (Carboplatin + Paclitaxel+Placebo): Patients receive paclitaxel and carboplatin as in arm I. Patients also receive oral placebo twice daily on days 2-19.
Arm/Group | Arm I (Carboplatin + Paclitaxel + Sorafenib) | Arm II (Carboplatin + Paclitaxel+Placebo)
Number analyzed (Participants) | 410 | 413
months | 11.1 [10.3 to 12.3] | 11.3 [9.8 to 12.2]
Statistical Analysis 1: Comparison: Arm I (Carboplatin + Paclitaxel + Sorafenib) vs Arm II (Carboplatin + Paclitaxel+Placebo); Test type: Superiority or Other; p = 0.863, Log Rank; Stratified log rank test is used for overall survival comparison, stratified on AJCC stage, ECOG Performance status and prior therapy status; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.87 to 1.18] — Arm II is the reference group

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as time from study entry to disease progression or death from any cause, whichever occurred first. Patients without disease progression were censored at last date of assessment. Disease progression was assessed by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0.
Time Frame: Tumor response was assessed after every 2 cycles during cycle 1 through 10, and every 3 cycles after cycle 10. Survival was assessed every 3 months if patient is < 2 years from study entry, and every 6 months if 2-5 years from study entry.
Population: Intention-to-treat population, n=821, two patients had no information about date of progression, and were excluded from the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Carboplatin + Paclitaxel + Sorafenib) | Arm II (Carboplatin + Paclitaxel+Placebo)
Number analyzed (Participants) | 409 | 412
months | 4.9 [4.5 to 5.6] | 4.2 [3.4 to 4.7]
Statistical Analysis 1: Comparison: Arm I (Carboplatin + Paclitaxel + Sorafenib) vs Arm II (Carboplatin + Paclitaxel+Placebo); Test type: Superiority or Other; p = 0.092, Log Rank — priori threshold for statistical significance: P<0.05; Stratified log rank test is used for progression-free survival comparison, stratified on AJCC stage, ECOG Performance status and prior therapy status; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.78 to 1.03] — Arm II is the reference group

3. Secondary Outcome: Objective Response (Complete and Partial Response) Rate
Description: Tumor response was assessed by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0. Objective response =complete response (CR) + partial response (PR). Complete response is defined as disappearance of all target lesions. Partial response is defined as at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum of longest diameters.
Time Frame: Tumor response was assessed after every 2 cycles during cycle 1 through 10. After cycle 10, tumor response was assessed after every 3 cycles.
Population: Intention-to-treat population, n=823
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Arm I (Carboplatin + Paclitaxel + Sorafenib) | Arm II (Carboplatin + Paclitaxel+Placebo)
Number analyzed (Participants) | 410 | 413
proportion | 0.205 [0.167 to 0.247] | 0.182 [0.146 to 0.222]
Statistical Analysis 1: Comparison: Arm I (Carboplatin + Paclitaxel + Sorafenib) vs Arm II (Carboplatin + Paclitaxel+Placebo); Test type: Superiority or Other; p = 0.427, Fisher Exact — priori threshold for statistical significance: P<0.05

ADVERSE EVENTS:
Time Frame: assessed at the end of each cycle (1 cycle = 3 weeks) while on study and for 30 days after the end of treatment
Arm/Group | Arm I (Carboplatin + Paclitaxel + Sorafenib) | Arm II (Carboplatin + Paclitaxel+Placebo)
Serious Adverse Events (participants affected / at risk) | 332/393 | 311/397
Other Adverse Events (participants affected / at risk) | 385/393 | 384/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Carboplatin + Paclitaxel + Sorafenib) (N=393) | Arm II (Carboplatin + Paclitaxel+Placebo) (N=397)
Allergic reaction (Immune system disorders) | 20 | 11
Otitis, middle ear (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 30 | 28
Hemolysis (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Investigations) | 108 | 91
Lymphopenia (Investigations) | 21 | 17
Neutropenia (Investigations) | 192 | 195
Thrombocytopenia (Investigations) | 92 | 35
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrial flutter (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
PVCs (Cardiac disorders) | 1 | 0
Cardiac-ischemia (Cardiac disorders) | 4 | 1
Hypertension (Vascular disorders) | 18 | 5
Hypotension (Vascular disorders) | 11 | 5
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 2
cardiac-other (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 63 | 56
Fever w/o neutropenia (General disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 3
Rigors/chills (General disorders) | 0 | 2
Weight loss (Investigations) | 2 | 1
INR increased (Investigations) | 1 | 0
activated partial thromboplastin time (PTT) (Investigations) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 13 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 58 | 8
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 | 0
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 47 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Death - multiorgan failure (General disorders) | 1 | 0
Death - sudden death (General disorders) | 2 | 1
Hot flashes (Vascular disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 21 | 9
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 21 | 19
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 29 | 15
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Muco/stomatitis (symptom) oral (Gastrointestinal disorders) | 2 | 1
Muco/stomatitis (symptom) stomach (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 16 | 11
Obstruction, small bowel NOS (Gastrointestinal disorders) | 1 | 2
Perforation, colon (Gastrointestinal disorders) | 2 | 1
Ulcer, duodenum (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 13 | 11
Gastrointestinal disorder-other (Gastrointestinal disorders) | 2 | 0
Hematoma (Vascular disorders) | 1 | 0
CNS, hemorrhage (Nervous system disorders) | 1 | 1
Abdomen, hemorrhage NOS (Gastrointestinal disorders) | 0 | 1
Colon, hemorrhage (Gastrointestinal disorders) | 1 | 1
Duodenum, hemorrhage (Gastrointestinal disorders) | 2 | 1
Lower GI, hemorrhage NOS (Gastrointestinal disorders) | 1 | 0
Stomach, hemorrhage (Gastrointestinal disorders) | 1 | 0
Kidney, hemorrhage (Renal and urinary disorders) | 1 | 0
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemorrhage-other (Vascular disorders) | 1 | 0
Colitis, infectious (e.g. C.diff) (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 24 | 17
Infection w/ gr304 neut, anal/perianal (Infections and infestations) | 0 | 1
Infection w/ gr304 neut, bladder (Infections and infestations) | 0 | 1
Infection w/ gr304 neut, bronchus (Infections and infestations) | 1 | 0
Infection w/ gr304 neut, catheter relate (Infections and infestations) | 1 | 0
Infection w/ gr304 neut, lung (Infections and infestations) | 2 | 2
Infection w/ gr304 neut, oral cavity (Infections and infestations) | 0 | 2
Infection w/ gr304 neut, pharynx (Infections and infestations) | 0 | 2
Infection w/ gr304 neut, skin (Infections and infestations) | 2 | 2
Infection w/ gr304 neut, upper airway (Infections and infestations) | 0 | 1
Infection w/ gr304 neut, urinary tract (Infections and infestations) | 4 | 1
Infection Gr002 neut, catheter (Infections and infestations) | 0 | 1
Infection Gr002 neut, colon (Infections and infestations) | 0 | 1
Infection Gr002 neut, foreign body (Infections and infestations) | 1 | 0
Infection Gr002 neut, lung (Infections and infestations) | 3 | 3
Infection Gr002 neut, pharynx (Infections and infestations) | 1 | 0
Infection Gr002 neut, skin (Infections and infestations) | 2 | 4
Infection Gr002 neut, soft tissue (Infections and infestations) | 0 | 1
Infection Gr002 neut, urinary tract (Infections and infestations) | 1 | 1
Infection Gr002 neut, wound (Infections and infestations) | 1 | 0
Infection w/ unk ANC lung (Infections and infestations) | 0 | 2
Infection w/ unk ANC mucosa (Infections and infestations) | 0 | 1
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 1 | 0
Opportunistic infection (Infections and infestations) | 1 | 1
Infection w/ gr304 neut, blood (Infections and infestations) | 9 | 9
Infection Gr002 neut, blood (Infections and infestations) | 1 | 1
Infection w/ unk ANC blood (Infections and infestations) | 0 | 1
Infection- other (Infections and infestations) | 2 | 1
Edema limb (General disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 4
Alkaline phosphatase increased (Investigations) | 5 | 3
Alkalosis (Metabolism and nutrition disorders) | 0 | 1
ALT, SGPT (Investigations) | 5 | 2
Serum amylase increased (Investigations) | 4 | 2
AST, SGOT (Investigations) | 3 | 2
Blood bilirubin increased (Investigations) | 3 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 3
Creatinine increased (Investigations) | 3 | 2
GGT increased (Investigations) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 17 | 19
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 12 | 11
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic/Laboratory-other (Investigations) | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint-function (Musculoskeletal and connective tissue disorders) | 1 | 0
Nonneuropathic lower extr muscle (Musculoskeletal and connective tissue disorders) | 5 | 0
Nonneuropathic upper extr muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 7 | 3
Ataxia (Nervous system disorders) | 1 | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 3 | 1
Dizziness (Nervous system disorders) | 2 | 8
Encephalopathy (Nervous system disorders) | 1 | 1
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 3
Depression (Psychiatric disorders) | 0 | 1
Neuropathy- motor (Nervous system disorders) | 12 | 10
Neuropathy- sensory (Nervous system disorders) | 81 | 59
Personality (Psychiatric disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 3
Cataract (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Vision photophobia (Eye disorders) | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 11 | 3
Bone, pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Cardiac/heart, pain (Cardiac disorders) | 1 | 1
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Chest/thoracic pain NOS (General disorders) | 1 | 2
Extremity limb, pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Head/headache (Nervous system disorders) | 2 | 2
Joint, pain (Musculoskeletal and connective tissue disorders) | 14 | 14
Lymph node, pain (Blood and lymphatic system disorders) | 1 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 18 | 22
Neuropathic, pain (Nervous system disorders) | 1 | 0
Pain NOS (General disorders) | 0 | 1
Pericardium, pain (General disorders) | 0 | 1
Pleura, pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin, pain (Skin and subcutaneous tissue disorders) | 1 | 0
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain-other (General disorders) | 2 | 1
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 6
Thrombosis/thrombus/embolism (Vascular disorders) | 4 | 8
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 1
Lipase increased (Investigations) | 14 | 6
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 21 | 9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Carboplatin + Paclitaxel + Sorafenib) (N=393) | Arm II (Carboplatin + Paclitaxel+Placebo) (N=397)
Anemia (Blood and lymphatic system disorders) | 191 | 195
Leukopenia (Investigations) | 135 | 146
Lymphopenia (Investigations) | 38 | 29
Neutropenia (Investigations) | 101 | 117
Thrombocytopenia (Investigations) | 182 | 131
Hypertension (Vascular disorders) | 87 | 38
Fatigue (General disorders) | 311 | 296
Fever w/o neutropenia (General disorders) | 19 | 25
Insomnia (Psychiatric disorders) | 47 | 39
Rigors/chills (General disorders) | 34 | 21
Sweating (General disorders) | 23 | 12
Weight loss (Investigations) | 62 | 25
Dry skin (Skin and subcutaneous tissue disorders) | 38 | 10
Flushing (Skin and subcutaneous tissue disorders) | 21 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 202 | 209
Pruritus/itching (Skin and subcutaneous tissue disorders) | 110 | 59
Rash/desquamation (Skin and subcutaneous tissue disorders) | 198 | 105
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 119 | 28
Skin-other (Skin and subcutaneous tissue disorders) | 20 | 7
Anorexia (Metabolism and nutrition disorders) | 137 | 118
Constipation (Gastrointestinal disorders) | 101 | 86
Dehydration (Metabolism and nutrition disorders) | 23 | 20
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 200 | 113
Dyspepsia (Gastrointestinal disorders) | 36 | 35
Muco/stomatitis (symptom) stomach (Gastrointestinal disorders) | 84 | 44
Nausea (Gastrointestinal disorders) | 206 | 230
Taste disturbance (Gastrointestinal disorders) | 57 | 54
Vomiting (Gastrointestinal disorders) | 104 | 117
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 21 | 5
Edema limb (General disorders) | 35 | 31
Hypoalbuminemia (Metabolism and nutrition disorders) | 36 | 27
Alkaline phosphatase increased (Investigations) | 46 | 29
Alanine aminotransferase (ALT, SGPT) (Investigations) | 48 | 33
Aspartate aminotransferase (AST, SGOT) (Investigations) | 56 | 29
Hyperglycemia (Metabolism and nutrition disorders) | 58 | 44
Lipase increased (Investigations) | 27 | 14
Hypomagnesemia (Metabolism and nutrition disorders) | 33 | 29
Hypokalemia (Metabolism and nutrition disorders) | 49 | 20
Hyponatremia (Metabolism and nutrition disorders) | 51 | 37
Metabolic/Laboratory-other (Metabolism and nutrition disorders) | 26 | 14
Dizziness (Nervous system disorders) | 52 | 45
Neuropathy-sensory (Nervous system disorders) | 262 | 265
Abdomen, pain (Gastrointestinal disorders) | 30 | 21
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 23 | 19
Head/headache (Nervous system disorders) | 46 | 34
Joint, pain (Musculoskeletal and connective tissue disorders) | 157 | 151
Muscle, pain (Musculoskeletal and connective tissue disorders) | 158 | 182
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 18
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 65 | 54
Hypocalcemia (Metabolism and nutrition disorders) | 37 | 17
Creatinine increased (Investigations) | 21 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less